CLINICAL TRIAL: NCT05203627
Title: Telehealth Intervention for Self-Management of Dietary Quality of Life After Gastric Cancer Surgery
Brief Title: Telehealth for the Self-Management of Dietary Quality of Life in Patients After Stomach Cancer Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19220; NCI-2021-12909 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19220 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-12-06; First posted 2022-01-24 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Gastric Carcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (telehealth session, guidebook) (Experimental): Patients receive 4 telehealth sessions over 1 hour each over 4 months. Patients also receive an intervention guidebook.
  Interventions: Other: Questionnaire Administration; Other: Telemedicine Visit
- Arm II (standard nutritional support) (Active Comparator): Patients receive standard nutritional support.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard nutritional support
  Other Names: standard of care; standard therapy
  Arms: Arm II (standard nutritional support)
Other: Questionnaire Administration — Ancillary studies
Other: Telemedicine Visit — Receive telehealth sessions
  Arms: Arm I (telehealth session, guidebook)

SUMMARY:
This clinical trial test whether taking part in a diet support intervention will help with patients nutrition and quality of life after surgery for esophagus or stomach cancer. The information learned by doing this research study may help patients get more information and/or support on eating after esophagus and stomach cancer surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the feasibility, retention, and satisfaction of the Telehealth Intervention for Self-Management of Eating after Gastric Surgery (TIMES) intervention as measured by the percentage of patients who a) agree to participate; b) complete a majority of the intervention (at least 2 sessions); and c) report satisfaction with the intervention (through structured exit interviews).

II. Assess the preliminary efficacy of TIMES for patient reported outcomes for quality of life (QOL), dietary symptoms, and self-management.

III. Assess the preliminary efficacy of TIMES for objective measures of patient nutrition.

OUTLINE: Patients are randomized in to 1 of 2 arms.

ARM I: Patients receive 4 telehealth sessions over 1 hour each over 4 months. Patients also receive an intervention guidebook.

ARM II: Patients receive standard nutritional support.

After completion of study, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* The ability to understand English or Spanish.
* Undergone curative intent surgery for gastric or gastroesophageal (GE) junction cancer.
* Began oral intake within the past month.
* Aged 21 years and older.
* Able to participate in telehealth sessions.
* This study will be conducted in patients aged 21 years or older who have undergone curative intent surgery for gastric or GE junction cancer.
* Age criterion for this trial is based on the National Institute of Health (NIH')s age criteria, which defines an adult as individuals aged 21 years and over. There are no restrictions related to performance status or life expectancy.
* All subjects must have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Telehealth Intervention - Percent Participation | Up to 6 months
  Feasibility of the Telehealth Intervention for Self-Management of Eating after Gastric Surgery (TIMES) intervention will be measured by the percentage of patients who agree to participate.
Feasibility of the Telehealth Intervention - Percent Completion | Up to 6 months
  Feasibility of the Telehealth Intervention for Self-Management of Eating after Gastric Surgery (TIMES) intervention will be measured by the percentage of patients who completes two sessions.
Retention of the TIMES intervention | Up to 6 months
  Measured by the percentage of patients who complete a majority of the intervention (at least 2 sessions).
Satisfaction of the TIMES intervention | Up to 6 months
  Measured by the percentage of patients who report satisfaction with the intervention (through structured exit interviews). Satisfaction and engagement will be assessed through the exit interview via qualitative data, content analysis approach.
Patient reported outcomes - European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ30): | Up to 6 months
  EORTC-QLQ30 will be assessed with a 30-item instrument for QOL assessment, with subscales/items for function, global health, general symptoms (fatigue, pain, nausea, and vomiting), and financial toxicity.
Patient reported outcomes - EORTC-Oesophago-Gastric Cancer Module | Up to 6 months
  (EORTC-OG25) will be assessed with a 25-item measure for esophagogastric cancer-specific symptoms and emotional well-being.
Patient reported outcomes - Patient Activation Measure (PAM) | Up to 6 months
  Patient Activation Measure (PAM) will be assessed by using a Guttman-like scale that reflects a patient's level of engagement and empowerment in their healthcare.
Patient reported outcomes - General Self-Efficacy Scale | Up to 6 months
  A General Self-Efficacy Scale developed by Jerusalem and colleagues contains 10 items that assess perceived confidence in self-management.
  Items are rated on a 4-point Likert scale.
Patient reported outcomes - The Post-Gastrectomy Nutrition Questionnaire | Up to 6 months
  The Post-Gastrectomy Nutrition Questionnaire is a tool developed by the investigators to assess patient knowledge about diet and nutrition after surgery for GE cancer.
  Each item addresses specific content discussed in the telehealth sessions to assess changes in knowledge. Scoring is based on the number of questions answered correctly.
Objective measures of patient nutrition - Weight | Up to 6 months
  Weight will be recorded at baseline and 6 months to examine the preliminary efficacy of the intervention on objective measures of patient nutrition. Weight will be measured by kg.
Objective measures of patient nutrition - Body Mass Index (BMI) | Up to 6 months
  Body Mass Index will be calculated and recorded by dividing weight in Kg by height in m^2 at baseline and 6 months to examine the preliminary efficacy of the intervention on objective measures of patient nutrition.
Objective measures of patient nutrition - Albumin levels | Up to 6 months
  Serum albumin levels collected as routine follow-up care will be recorded at baseline and 6 months to examine the preliminary efficacy of the intervention on objective measures of patient nutrition. Albumin level will be measured g/dl.
Objective measures of patient nutrition - Skeletal mass Index | Up to 6 months
  Sarcopenia/skeletal muscle mass will be calculated at baseline and 6 months through CT scans performed as part of routine follow-up for gastroesophageal cancer include cross-sectional images at the level of the third lumbar vertebra (L3). The cross-sectional area of skeletal muscle mass in this region has been found in multiple studies to correlate with total body skeletal muscle mass. Skeletal muscle mass will be quantified using well described techniques applying a predefined Hounsfield unit (HU) threshold of -25 to 150 HU for skeletal muscle mass. Muscle boundaries will be corrected manually when necessary to obtain cross-sectional areas (cm2) for skeletal muscle. Skeletal muscle index (SMI, cm2/m2) is defined as the cross-sectional area of muscle at the L3 level normalized for BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Y Kim, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States